CLINICAL TRIAL: NCT05878353
Title: Influence of Local Doxycycline on the Inflammatory Status of Intrabony Defects and Clinical Outcomes of Periodontal Regeneration: a Randomized Controlled Trial
Brief Title: Influence of Local Doxycycline on the Outcomes of Periodontal Regeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DoxyTurin
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subgingival instrumentation plus local doxycycline (Experimental): Gentle debridement plus local doxycycline administered 2 weeks prior to periodontal regeneration.
  Interventions: Procedure: Decontamination of the pocket with local doxycycline
- Subgingival instrumentation alone (Active Comparator): Gentle debridement alone performed 2 weeks prior to periodontal regeneration.
  Interventions: Procedure: Decontamination of the pocket with mechanical instrumentation

INTERVENTIONS:
Procedure: Decontamination of the pocket with local doxycycline — Gentle debridement will be performed under local anesthesia (mepivacain 2% 1:1000) for a time of 5 minutes by mean of ultrasonic devices by the same experienced clinician. Great attention will be made to avoid marginal and interproximal soft tissue damage. Local doxycycline was administered according to the manufacturer's instruction. Briefly, the plastic needle of the syringe will be inserted into the sulcus and the product will be progressively released in the periodontal pocket up to the gingival margin. The syringe will be then removed and a cotton pellet used to compact the gel into the sulcus. Patients will be then instructed not to floss or use interdental brushes in that area for the following 10 days.
  Arms: Subgingival instrumentation plus local doxycycline
Procedure: Decontamination of the pocket with mechanical instrumentation — Gentle debridement will be performed under local anesthesia (mepivacain 2% 1:1000) for a time of 5 minutes by mean of ultrasonic devices by the same experienced clinician. Great attention will be made to avoid marginal and interproximal soft tissue damage.
  Arms: Subgingival instrumentation alone

SUMMARY:
In this double-blinded randomized clinical trial, patients presenting periodontal intrabony defects requiring regenerative surgery and showing BoP will be included. Experimental sites at T-0 will be randomly treated with gentle debridement and administration of local DOX (test group) or with debridement alone (control group). After 2 weeks (T-1), defects will be treated by means of minimally invasive surgical technique. 14 days after the surgery (T-2) the EHI will be evaluated by a blinded examiner. Patients will be recalled each 2 months up to 12 months (T-3). At T-0, T-1 and T-3 periodontal examination and radiographic analysis will be done.

ELIGIBILITY:
Inclusion Criteria:

* 1) diagnosis of Stage III or IV periodontitis (Tonetti et al. 2018);
* 2) FMPS and FMBS < 15% at the time of enrollment;
* 3) etiological periodontal therapy completed at least 3 months prior to screening;
* 4) presence of one natural tooth having a vertical defect with residual PPD ≥ 6 mm and a radiographic intrabony component ≥ 3 mm and BoP + requiring periodontal regenerative surgery.

Exclusion Criteria:

* 1) age < 18 years;
* 2) smoking habits (> 10 cigarettes/day);
* 3) contraindications for periodontal surgery;
* 4) systemic diseases affecting periodontal healing;
* 5) pregnancy and lactation;
* 6) history of periodontal surgery at the experimental teeth;
* 7) allergies to doxycycline and tetracyclines;
* 8) assumption of antibiotics in the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level change | 12 months
  Clinical attachment level will be assessed on the experimental teeth using periodontal probe (PCP 15/11.5, Hu-Friedy, Chicago, IL, USA)

SECONDARY OUTCOMES:
Radiographic bone level change | 12 months
  Periapical standardized radiographs will be taken by a clinician masked to the clinical measurements using the paralleling technique and individually customized bite-blocks (RINN XCP Film Holding Instruments, Dentsply, York, USA)
Probing pocket depth change | 12 months
  Probing depth will be assessed on the experimental teeth using periodontal probe (PCP 15/11.5, Hu-Friedy, Chicago, IL, USA)
Bleeding on probing reduction | 12 months
  Bleeding on probing will be assessed on the experimental teeth using periodontal probe (PCP 15/11.5, Hu-Friedy, Chicago, IL, USA)

CONTACTS AND LOCATIONS:
Locations (1):
- CIR Dental School, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aimetti M, Baima G, Lorenzetti V, Aliyeva N, Bottone M, Mariani GM, Romano F. A BiO-Optimizing Site Targeted (BOOST) Approach to Periodontal Regeneration Through Local Doxycycline Prior to Surgery: A Randomized Clinical Trial. J Periodontal Res. 2025 Jan 27. doi: 10.1111/jre.13389. Online ahead of print. PMID 39868481